CLINICAL TRIAL: NCT00634205
Title: A Phase II Study Assessing the Activity of Valproate Acid Plus Doxorubicin in Refractory or Recurrent Malignant Mesothelioma
Brief Title: Phase II Study of Valproate and Doxorubicin in Malignant Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Lung Cancer Working Party (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELCWP-01062
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Malignant Mesothelioma
Keywords: Mesothelioma; Valproate; Doxorubicin; Chemotherapy; Phase II
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma | interventions — Valproic Acid; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Continuous oral administration of valproate plus every 3 weeks, intravenous administration of doxorubicin
  Interventions: Drug: Valproate plus doxorubicin

INTERVENTIONS:
Drug: Valproate plus doxorubicin — Valproate 20-30 mg/kg orally (in order to obtain serum concentration between 50-100 mcg/ml) Doxorubicin 60 mg/m² intravenously every 3 weeks

SUMMARY:
The purpose of this study is to determine the response rate to the combination of doxorubicin and valproate acid in patients with MM failing after at least one previous chemotherapy regimen including platinum derivatives .

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of malignant mesothelioma
* Unresectable or inoperable malignant mesothelioma failing after at least one prior chemotherapy regimen including platinum derivatives (cisplatin or carboplatin)
* At least one evaluable or measurable CT-lesion
* Availability for participating in the detailed follow-up of the protocol
* Signed informed consent

Exclusion Criteria:

* Patients who are candidates for surgery with curative intent
* Patient who were previously treated with anthracyclin derivatives
* Performance status < 60 on the Karnofsky scale
* A history of prior malignant tumour, except non-melanoma skin cancer or in situ carcinoma of the cervix and cured malignant tumour (more than 5-year disease free interval)
* A history of prior HIV infection
* Polynuclear cells < 2,000/mm³
* Platelet cells < 100,000/mm³
* Abnormal coagulation tests (aPTT, PTT, prothrombin time) and/or decreased fibrinogen
* Serum bilirubin >1.5 mg/100 ml
* Transaminases more than twice the normal range
* Serum creatinine > 1.5 mg/100 ml
* Recent myocardial infarction (less than 3 months prior to date of diagnosis)
* Congestive cardiac failure (ejectional fraction of the left ventricle < 50%) or uncontrolled cardiac arrhythmia
* Uncontrolled infectious disease
* Active epilepsy needing a specific treatment
* Concomitant treatment with IMAO, carbamazepine, mefloquine, phenobarbital, primidone, phenytoïn, lamotrigine, zidovudine
* Pregnancy or refusal to use active contraception
* A known allergy to valproate acid and/or doxorubicin
* Serious medical or psychological factors which may prevent adherence to the treatment schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-07; Primary Completion 2009-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Response rate | Every 3 courses

SECONDARY OUTCOMES:
Survival | Survival will be dated from the day of registration until death or last follow up
Toxicity | After each course of chemotherapy and at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Berghmans, MD, Study Chair — European Lung Cancer Working Party
Locations (8):
- Belgium (7):
  - Department of Pneumology CHR St joseph - Warquignies, Boussu
  - Department of Intensive Care Unit and Thoracic Oncology Institut Jules Bordet, Brussels
  - Department of Pneumology Hôpital Ixelles-Molière, Brussels
  - Department of Pneumology CHU Charleroi, Charleroi
  - Department of Pneumology Hôpital Saint-Joseph, Gilly
  - Hôpital Ambroise Paré, Mons
  - CH Peltzer-La Tourelle, Verviers
- Department of Pneumology CHRU Lille, Lille, France

REFERENCES:
- [Derived] Scherpereel A, Berghmans T, Lafitte JJ, Colinet B, Richez M, Bonduelle Y, Meert AP, Dhalluin X, Leclercq N, Paesmans M, Willems L, Sculier JP; European Lung Cancer Working Party (ELCWP). Valproate-doxorubicin: promising therapy for progressing mesothelioma. A phase II study. Eur Respir J. 2011 Jan;37(1):129-35. doi: 10.1183/09031936.00037310. Epub 2010 Jun 7. PMID 20530048
- See also: Click here for more information on the protocol — http://www.elcwp.org
- See also: Trials registry of the French National Cancer Institute — http://www.e-cancer.fr